CLINICAL TRIAL: NCT01516203
Title: Randomized, Open Label, Multiple Dose Phase 2a Study of the Early Bactericidal Activity of AZD5847 in Adults With Pulmonary Tuberculosis
Brief Title: Phase 2a EBA Trial of AZD5847
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0006
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2014-03-19

CONDITIONS: Tuberculosis
Keywords: AZD5847; dose-ranging; Mycobacterium tuberculosis; Rifafour; tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — posizolid; Ethambutol; Isoniazid; Pyrazinamide; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1 (Experimental): AZD5847 500 mg orally once daily given to 15 male and female subjects aged 18 to 65 years with newly diagnosed sputum smear positive pulmonary tuberculosis
  Interventions: Drug: AZD5847
- Arm 2 (Experimental): AZD5847 500 mg orally twice daily given to 15 male and female subjects aged 18 to 65 years with newly diagnosed sputum smear positive pulmonary tuberculosis
  Interventions: Drug: AZD5847
- Arm 3 (Experimental): AZD5847 1200 mg orally once daily given to 15 male and female subjects aged 18 to 65 years with newly diagnosed sputum smear positive pulmonary tuberculosis
  Interventions: Drug: AZD5847
- Arm 4 (Experimental): AZD5847 800 mg orally twice daily given to 15 male and female subjects aged 18 to 65 years with newly diagnosed sputum smear positive pulmonary tuberculosis
  Interventions: Drug: AZD5847
- Arm 5 (Active Comparator): Rifafour e-275 mg tablets given to 15 male and female subjects aged 18 to 65 years with newly diagnosed sputum smear positive pulmonary tuberculosis
  Interventions: Drug: Ethambutol, isoniazid, pyrazinamide, rifampin

INTERVENTIONS:
Drug: AZD5847 — Eligible subjects will be randomly assigned to receive monotherapy with one of four doses of oral AZD5847 for 14 days: 500 mg orally once daily, 500 mg orally twice daily, 1200 mg orally once daily, or 800 mg orally twice daily.
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: Ethambutol, isoniazid, pyrazinamide, rifampin — Eligible subjects will be randomly assigned to receive treatment with standard 4 drug anti-tuberculosis regimen: Rifafour e-275 mg tablets (75 mg isoniazid/150 mg Rifampin/275 mg Ethambutol/400 mg Pyrazinamide) orally, dosed by body weight for 14 days.
  Arms: Arm 5

SUMMARY:
The purpose of this study is to assess the early bacterial activity (EBA) from day 0 to day 14 of Astra Zeneca Drug (AZD5847) at four different doses and schedules (500 mg once daily, 500 mg twice daily, 1200 mg once daily, and 800 mg twice daily) in subjects with newly-diagnosed sputum smear positive pulmonary TB. A total of 75 subjects will be enrolled, with 15 randomized to each AZD5847 study arm or standard treatment with Rifafour. Duration of drug treatment is 14 days.

DETAILED DESCRIPTION:
This is a study of early bactericidal activity (EBA) in treatment-naïve patients with active pulmonary tuberculosis. This prospective, randomized, open-label study that will compare the effect of monotherapy with each of four dose levels of AZD5847 to that of an active control (Rifafour administered orally once daily) on the concentration of Mycobacterium tuberculosis (M. tb) in expectorated sputum (colony-forming units per mL of sputum). Daily quantitative sputum cultures will be performed during treatment and analyzed by investigators who will be blinded to the assigned treatment. The duration of therapy will be 14 days in order to support an assessment of early bactericidal activity (days 0-2) and sterilizing activity (days 3-14). Because of the risk of emergence of drug resistance in TB patients treated with a single active drug, regulatory and ethical requirements restrict monotherapy to a maximum duration of 14 days (EMEA Draft TB Guidance 2008). The study will utilize a standard design and will thus support comparison with other marketed and investigational antimycobacterial agents (Donald and Diacon 2008). The primary aim of the study is to assess the EBA 0-14 of AZD5847 at four different doses and schedules (500 mg once daily, 500 mg twice daily, 1200 mg once daily, and 800 mg twice daily) in subjects with newly-diagnosed sputum smear positive pulmonary TB. The secondary aim is to assess the EBA 0-2 and EBA 2-14 of AZD5847 at the above doses.

ELIGIBILITY:
Inclusion Criteria:

- Adults, male or female, age 18 to 65 years - Post-menopausal women under the age of 65 years will be included in the study. Women of childbearing potential must be using or agree to use an adequate method of birth control through the end of study follow up. These methods include: total sexual abstinence; a single male partner who has been vasectomized combined with use of a condom; a combination of two effective birth control methods from the following list: a. an intrauterine device plus a condom; b. a tubal ligation (tubes tied) plus a condom; c. Depo-provera injections plus a condom; d. Intravaginal ring plus a condom - Newly diagnosed sputum smear-positive pulmonary tuberculosis as confirmed by at least one sputum AFB + smear (at least grade 1+ using the WHO/IUATLD grading scale) - Willing and able to provide informed consent - Hemoglobin >/= 8 gm/dL - Serum creatinine < 2 mg/dL (<176.8 umol/L) - Serum AST < 3.0 times the upper limit of normal for the testing laboratory and total bilirubin < 1.3 mg/dL - Random blood glucose < 150 mg/dL (< 8.32 mmol/L) - If HIV-positive, not currently on ART, CD4 count> 350 muL^-1 and/or no need to start ART in the opinion of the local investigator - Cough productive of at least 10 ml (two teaspoons) of sputum daily per patient report over the week prior to enrollment. - Chest radiograph compatible with pulmonary TB. - Negative sputum Xpert™ MTB/RIF test for rifampin resistance. - Negative urine pregnancy test

Exclusion Criteria:

- HIV infection with CD4 count of </=350muL^-1 and/or the need to start ART in the opinion of the local investigator. - Weight less than 40 kg or greater than 90 kg - Presence of hemoptysis. Subjects who cough up frank blood (more than blood streaked sputum) will not be eligible for enrollment. - Subjects with rifampin resistance as determined by the Xpert test as screening. - Pregnant or breastfeeding women - Presence of pneumothorax on pretreatment chest radiograph - Clinical suspicion of disseminated tuberculosis or tuberculous meningitis or pulmonary TB requiring immediate start of standard chemotherapy in the opinion of the local investigator - Presence of serious underlying medical illness, such as liver failure, renal failure,any diabetes mellitus, chronic alcoholism (> 3 alcoholic drinks per day), decompensated heart failure, cardiac arrhythmias, hematologic malignancy or subjects receiving myelosuppressive chemotherapy. - Allergy or contraindication to study drugs - Prior treatment for TB with antituberculous medications (isoniazid, rifampin, pyrazinamide, ethambutol or streptomycin or those treated with other antibiotics with known activity against MTB during the preceding 6 months (for example aminoglycosides, fluoroquinolones, carbapenems and linezolid) - Subjects taking monoamine oxidase (MAO) inhibitors or selective serotonin release inhibitor (SSRI) medications - Total white blood cell count less than 3000/mm^3 - Platelet count less than 150,000/mm^3 - Subjects with QTcF> 450 msec, QTcF < 340 msec, and/or family history of long QT syndrome - Subjects unlikely in the opinion of the local investigator to be able to comply with the requirements of the study protocol - Subjects whose urine tests positive for INH metabolites, indicating they are already receiving anti-TB treatment. - History of tuberculosis less than 5 years ago, history of more than one episode of tuberculosis, history of drug resistant tuberculosis, or household contact with an individual who has confirmed drug-resistant tuberculosis. - Known arrhythmias or other cardiac conditions - Active severe dermatologic disease (Grade 3 or Grade 4 per DMID Adult Toxicity Table) - Immunosuppressive conditions or receiving immunosuppressive medications - A history of optic neuritis. - Subjects on antiretroviral therapy for HIV (including AZT, 3TC, FTC, D4T, ddI, ddC, tenofovir, abacavir, nevirapine, efavirenz, ritonavir, lopinavir, atazanavir, saquinavir, darunavir, indinavir, raltegravir) - Subjects taking drugs capable of prolonging the QTc interval, such as type Ia and III anti-arrhythmics - Random urine toxicology screen positive for cocaine or methamphetamines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2013-12-12 (Actual); Study Completion 2013-12-24 (Actual)

PRIMARY OUTCOMES:
Early Bactericidal Activity: Rate of change in sputum colony forming unit (CFU) counts (bactericidal activity) during the entire 14 days of study drug administration (EBA0-14) | Day 0 to Day 14

SECONDARY OUTCOMES:
Adverse event collection: Complete blood count, coagulation panels, liver function tests, Creatine phosphokinase, urinalysis and 12-lead electrocardiograms as well as unsolicited events (adverse events, serious adverse events). | Day 0 to Day 28
Change in Mycobacterium tuberculosis (MTB) mRNA in sputum by RT-PCR for fbpB, hspX, icl1, rrnA-p1 and other specific mycobacterial mRNA targets of interest over the periods (baseline and Days 2, 4, 8, 14) | Baseline and Days 2, 4, 8, 14
Change in urine, sputum, and serum metabolomic biomarkers over the periods (baseline and Days 8, 14) | Baseline and Days 8, 14
Pharmacokinetic and pharmacodynamic parameters Tmax, Cmax, half life, AUC, AUC/MIC, Cmax, Cmax/MIC, time > MIC using non-compartmental analysis, compartmental and population models | Day 1, 3, 5, 10 and 14
Rate of change in sputum CFU counts (bactericidal activity) during the first 2 days of study drug administration (traditional EBA; EBA0-2) | Day 0 to Day 2
Rate of change in sputum CFU counts (bactericidal activity) during the first 2 to 14 days of study drug administration (traditional EBA; EBA2-14) | Day 2 to Day 14
The change in time after inoculation until culture detection (time to detection; TTD) in MGIT enriched liquid culture media over the period Day 0 to Day 2 | Day 0 to Day 2
The change in time after inoculation until culture detection (time to detection; TTD) in MGIT enriched liquid culture media over the period Day 2 to Day 14 | Day 2 to Day 14
The change in time after inoculation until culture detection (time to detection; TTD) in Mycobacterial Growth Indicator Tube (MGIT) enriched liquid culture media over the period Day 0 to Day 14 | Day 0 to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Task Clinical Research Centre, Ekurhuleni, Gauteng, South Africa

REFERENCES:
- [Result] Alsultan A, Furin JJ, Du Bois J, van Brakel E, Chheng P, Venter A, Thiel B, Debanne SA, Boom WH, Diacon AH, Johnson JL, Peloquin CA. Population Pharmacokinetics of AZD-5847 in Adults with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e01066-17. doi: 10.1128/AAC.01066-17. Print 2017 Oct. PMID 28739794
- [Result] Furin JJ, Du Bois J, van Brakel E, Chheng P, Venter A, Peloquin CA, Alsultan A, Thiel BA, Debanne SM, Boom WH, Diacon AH, Johnson JL. Early Bactericidal Activity of AZD5847 in Patients with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6591-6599. doi: 10.1128/AAC.01163-16. Print 2016 Nov. PMID 27550361